CLINICAL TRIAL: NCT03604523
Title: Effectiveness of Semi-rigid Savary Dilators vs. Balloon Dilators During Esophageal Dilation in the Treatment of Esophageal Dysmotility
Brief Title: Esophageal Dysmotility - Prospective Study Evaluating Methods for Esophageal Dilation
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Slow enrollment
Sponsor: University of Massachusetts, Worcester (Other)
Responsible Party: Principal Investigator, David Cave, Professor, University of Massachusetts, Worcester
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: H00004174
Record Dates: First submitted 2018-06-26; First posted 2018-07-27 (Actual); Results first posted 2021-04-13 (Actual); Last update posted 2021-04-13 (Actual); Status verified 2021-03

CONDITIONS: Esophageal Dysmotility
MeSH Terms: conditions — Esophageal Motility Disorders

STUDY DESIGN:
Intervention Model Description: Participants are randomized to procedure, but if participant fails the first procedure they are given the opportunity to crossover to the other arm for a follow up procedure.
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

ARMS (2):
- Dilation by Balloon (Active Comparator): Esophageal dilation by balloon device.
  Interventions: Device: Dilation by Balloon
- Dilation by Semi-rigid Savary (Active Comparator): Esophageal dilation by semi-rigid savary device.
  Interventions: Device: Dilation by Semi-rigid Savary

INTERVENTIONS:
Device: Dilation by Balloon — Esophageal dilation by balloon device.
  Arms: Dilation by Balloon
Device: Dilation by Semi-rigid Savary — Esophageal dilation by semi-rigid savary device
  Arms: Dilation by Semi-rigid Savary

SUMMARY:
The purpose of the study is to prospectively evaluate the most effective treatment of esophageal dysmotility that alleviates symptoms of dysphagia and improves quality of life.

Current practice uses either semi-rigid Savary dilators or balloon dilators for esophageal dilation to treat dysphagia due to esophageal dysmotility. The study aims to show which treatment method is more effective in alleviating symptoms, since there are no other treatments available. The null hypothesis is that there is no difference between the clinical benefits of each treatment.

DETAILED DESCRIPTION:
Both the Savary and balloon dilators are used as routine procedure at University of Massachusetts (UMass) Medical School's academic medical center UMass Memorial Health Care (UMMHC). Gastroenterologists are required as part of their training to be familiar with both types of procedures. This study aims to definitively determine which treatment method is more effective in alleviating the symptoms of esophageal dysmotility.

The primary clinical endpoint is to assess the therapeutic efficacy of different types of dilators in an esophageal dilation procedure in patients with esophageal dysmotility. This will be evaluated through the use of the dysphagia scale (Knyrim et al, 1993). The secondary aims are to assess time to relapse, diet improvement, as well as change in quality of life. Investigators will determine time to relapse by time between the dilation procedures. Participants are instructed to contact the GI office to schedule another dilation if they feel as though the therapeutic effect of the procedure has subsided and they are in need of additional relief. Diet will be assessed using the diet score (Cox et al, 1998) and quality of life will be assessed using the Short Form (SF) SF-12 Health Survey.

If patients fail the first procedure, they can be offered the alternative procedure at a later date. Both the patient and physician must agree that the treatment has not worked, and then the patient will be given the opportunity to cross over to the other procedure, still blinded to the device that will be used. Investigators will conduct an interim evaluation to assess the progress of the study and degree of crossover. This will ensure that all subjects are given the opportunity to have both devices used in the event that one is significantly superior to the other.

ELIGIBILITY:
Inclusion Criteria:

* > 18 years old
* Dysphagia to liquids and/or solids
* Diagnosis of esophageal dysmotility
* Normal endoscopic exam

Exclusion Criteria:

* Diagnosis of achalasia
* Defined strictures or webs
* Vulnerable populations:
* Adults unable to consent (Individuals who are not yet adults (infants, children, teenagers), Pregnant women, Prisoners)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Actual)
Dates: Start 2014-08-14 (Actual); Primary Completion 2016-11-26 (Actual); Study Completion 2016-11-26 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: David Cave, MD, Principal Investigator — Professor of Medicine, UMass Medical School
Locations (1):
- UMass Memorial Medical Center, Worcester, Massachusetts, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Dilation by Balloon | Dilation by Semi-rigid Savary
Started | 5 | 5
Completed | 4 | 5
Not Completed | 1 | 0
Not completed — Physician Decision | 1 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Dilation by Balloon | Dilation by Semi-rigid Savary | Total
Number analyzed (Participants) | 5 | 5 | 10
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 4 | 2 | 6
  >=65 years | 1 | 3 | 4
Age, Continuous [Mean (Full Range); unit: years] | 66 [52 to 78] | 56.8 [45 to 68] | 61.4 [45 to 78]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 4 | 4 | 8
  Male | 1 | 1 | 2
Region of Enrollment [Number; unit: participants]
  United States | 5 | 5 | 10

OUTCOME MEASURES:

1. Primary Outcome: Therapeutic Efficacy as Measured by Change in Dysphagia Scale Score
Description: Therapeutic efficacy of different types of dilators in an esophageal dilation procedure in patients with esophageal dysmotility. This will be evaluated through the use of the dysphagia scale (Knyrim 1993). Minimum score is 0. Maximum score is 4. Higher scores indicate a worse outcome. The data presented represent a change from baseline to 6 months calculated as the value at 6 months minus the value at baseline.
Time Frame: Baseline to 6 months post-procedure
Population: Data missing from participants who were lost to follow up at 6 months. Data provided for participants who completed 6 month follow up dysphagia score assessment.
Measure: Mean (Full Range); unit: units on a scale
Arm/Group | Dilation by Balloon | Dilation by Semi-rigid Savary
Number analyzed (Participants) | 3 | 4
units on a scale | -1 [-2 to 0] | -0.25 [-1 to 0]

2. Secondary Outcome: Participants With Relapse
Description: Participants who required esophageal dilation within time frame
Time Frame: Baseline to 6 months
Population: The population of those who were enrolled in the arms and received the assigned intervention.
Measure: Count of Participants; unit: Participants
Arm/Group | Dilation by Balloon | Dilation by Semi-rigid Savary
Number analyzed (Participants) | 4 | 5
Participants | 2 | 0

3. Secondary Outcome: Time to Relapse
Description: For the participants who relapsed, measure of time to relapse based on time from procedure to need for additional dilation due to subsidence of therapeutic effect of procedure.
Time Frame: Initial intervention to second dilation
Population: Participants who experienced a relapse in time period from baseline to 6 months. Only 2 participants in the dilation by balloon group experienced a relapse. This population was used to calculate the time to relapse. No participants in the dilation by semi-rigid Savary experienced a relapse during this time.
Measure: Mean (Full Range); unit: days
Arm/Group | Dilation by Balloon | Dilation by Semi-rigid Savary
Number analyzed (Participants) | 2 | 0
days | 72 [27 to 117] |

4. Secondary Outcome: Diet Dysphagia Score Change
Description: Diet dysphagia score change based on change to Cox diet score, taken from Table 1 of publication Gut, 1988, 29, 1741-1747. The scores are determined based on the foods that cause dysphagia. The minimum value on the score is 0 (no dysphagia), followed by 1 (dysphagia with meat), 2 (dysphagia with bread), 3 (dysphagia with semi-solids), 4 (dysphagia with liquids), and the maximum score is 5 (total dysphagia). A higher score indicates a worse clinical outcome. The data presented represent a change from baseline to 6 months calculated as the value at 6 months minus the value at baseline
Time Frame: baseline to 6 months post procedure
Population: Data is incomplete. Only 1 participant provided full diet score survey at 6 months.
Measure: Number; unit: units on a scale
Arm/Group | Dilation by Balloon | Dilation by Semi-rigid Savary
Number analyzed (Participants) | 1 | 0
units on a scale | -2 |

ADVERSE EVENTS:
Time Frame: Baseline to 6 months after procedure
Arm/Group | Dilation by Balloon | Dilation by Semi-rigid Savary
All-Cause Mortality (participants affected / at risk) | 0/4 | 0/5
Serious Adverse Events (participants affected / at risk) | 1/4 | 1/5
Other Adverse Events (participants affected / at risk) | 4/4 | 5/5
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Dilation by Balloon (N=4) | Dilation by Semi-rigid Savary (N=5)
Migraine (Nervous system disorders) | 1 (1) | 0 (0)
Shortness of breath (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Dilation by Balloon (N=4) | Dilation by Semi-rigid Savary (N=5)
Dysphagia (Gastrointestinal disorders) | 3 (3) | 0 (0)
Joint pain (Musculoskeletal and connective tissue disorders) | 2 (2) | 1 (1)
Chest pain (General disorders) | 1 (1) | 1 (1)
Leg cramps (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Leg pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Dyspepsia (Gastrointestinal disorders) | 0 (0) | 1 (1)

LIMITATIONS AND CAVEATS:
Recruitment was much slower than planned and the study was terminated early with only 15.6% of overall study goal enrolled. Early termination led to small numbers of subjects analyzed. Subjects unable to be reached for followup led to missing data for outcome measures.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes